CLINICAL TRIAL: NCT02112747
Title: Ohio Colorectal Cancer Prevention Initiative: Adherence to Colon Cancer Screening (ACCS) Project:Your Personal Prescription For Colorectal Cancer Screening.
Brief Title: Adherence to Colon Cancer Screening (ACCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-12230; NCI-2013-01146 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Colorectal Cancer Prevention; Colorectal Cancer Screening; ACCS; Lynch Syndrome; LS
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: website access only (No Intervention): There is no intervention with this arm. Completion of the website is part of enrollment.
- Arm 2: patient navigator (Experimental): The intervention consists of participants receiving the services of a patient navigator to address individual barriers to adhering to the "personal prescription" for colon and rectal cancer screening.
  Interventions: Other: Patient Navigator
- Arm 3: genetic counseling (No Intervention): There is no intervention in this arm. Patients diagnosed as positive for Lynch Syndrome use genetic counseling to discuss medical and family history and genetic risk of CRC, including genetic factors such as DNA mismatch repair genes, autosomal dominant inheritance, cancer risks associated with LS, screening recommendations, and genetic testing. There is no intervention. This is standard care.
- Arm 4:Gen. counselor & patient navigator (Experimental): Participants diagnosed positive for Lynch syndrome use genetic counseling as in Arm 3 and in addition receive the services of a patient navigator to address individual barriers to adhering to the CRC screening recommendations.
  Interventions: Other: Patient Navigator

INTERVENTIONS:
Other: Patient Navigator — Patients are randomized to receive the assistance of a patient navigator to understand, obtain assistance with following the screening recommendations of the personal prescription given to them by the website survey.
  Arms: Arm 2: patient navigator; Arm 4:Gen. counselor & patient navigator

SUMMARY:
This randomized clinical trial studies website access or genetic counseling with or without patient navigators on adherence to colorectal cancer screening recommendations in patients with newly diagnosed colorectal cancer and their first degree relatives. Websites for colorectal cancer prevention and genetic counseling may be effective methods to help people learn about cancer screening. Patient navigators may improve adherence to colorectal cancer screening recommendations. It is not yet known whether website access or genetic counseling is more effective with or without patient navigators.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the comparative-effectiveness of the interventions (i.e., website +/- navigator or genetic counseling +/- navigator) in a randomized controlled trial, using colorectal cancer (CRC) cases as the unit of randomization/analysis on adherence to individualized CRC screening recommendations.

SECONDARY OBJECTIVES:

I. Examine the cost effectiveness of the interventions, assessing the effect of the interventions on subgroups (i.e., Lynch syndrome positive vs. Lynch syndrome negative; probands vs. relatives; older vs. younger patients, etc), and barriers to adherence, as well as how the navigators resolve barriers.

II. Overscreening will be explored.

OUTLINE: Participants are assigned to 1 of 2 study components based on LS status. Within each component, participants are randomized to 1 of 2 arms.

COMPONENT #1 (Lynch Negative Proband and their first degree relatives (FDRs):

ARM I: Participants access a website to deliver a "personalized prescription for CRC prevention" based on age, Lynch Syndrome status, cancer history, age of 1st degree relative with CRC, and personal CRC screening history.

ARM II: Participants access a website as in Arm I and receive the services of a patient navigator to address individual barriers to adhering to the "personal prescription" within 1 month.

COMPONENT #2 (Lynch Positive Proband and their FDRs):

ARM III (Lynch positive proband): Participants use genetic counseling to discuss medical and family history and genetic risk of CRC, including genetic factors such as deoxyribonucleic acid (DNA) mismatch repair genes, autosomal dominant inheritance, cancer risks associated with LS, screening recommendations, and genetic testing.

ARM IV (Lynch positive proband): Participants use genetic counseling as in Arm III and receive the services of a patient navigator to address individual barriers to adhering to the CRC screening recommendations within 1 month.

After completion of study treatment, patients are followed up at 12-14 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with colorectal adenocarcinoma at Ohio State University (OSU) (or a participating Ohio hospital) with sufficient tumor available to perform the microsatellite instability (MSI) test, regardless of age at diagnosis or family history
* First-degree relatives of the cases who test positive for LS
* First-degree relatives of the cases who test negative for LS

Exclusion Criteria:

* Pregnant women
* Prisoners
* Individuals who are cognitively impaired

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1900 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Successfully following screening guidelines appropriate to the participant's risk profile | Up to 14 months
  For participants who are within the recommended guidelines, success would be defined as receiving no further screening. For those outside of the recommended guidelines, success would entail receiving a screening test. The outcome will combine medical record review and self-report by using medical record review when available and self-report otherwise. Evaluations will use a generalized estimating equations (GEE) approach with empirical sandwich variance estimators.

SECONDARY OUTCOMES:
Cost effectiveness of the interventions | Up to 14 months
  Analysis will consist of a cost analysis of the intervention incorporating project expenditures and both financial and non-financial costs incurred by the project participants. Financial benefits from the project will be incorporated into the cost analysis to produce a net cost of the interventions. These financial benefits will include expenditures for unnecessary or "overscreening" prevented by the interventions. The results of the net cost analysis will be combined with the outcome measures for screening interventions to establish the cost per guideline concordant screening.

CONTACTS AND LOCATIONS:
Overall Officials: Electra Paskett, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paskett ED, Bernardo BM, Young GS, Katz ML, Reiter PL, Tatum CM, Oliveri JM, DeGraffinreid CR, Gray DM, Pearlman R, Hampel H. Comparative Effectiveness of Two Interventions to Increase Colorectal Cancer Screening for Those at Increased Risk Based on Family History: Results of a Randomized Trial. Cancer Epidemiol Biomarkers Prev. 2020 Jan;29(1):3-9. doi: 10.1158/1055-9965.EPI-19-0797. Epub 2019 Oct 30. PMID 31666284
- See also: The Jamesline — http://cancer.osu.edu